CLINICAL TRIAL: NCT05740540
Title: Customizable Cooperative Multi-joint Control to Enhance Walking Mobility After Stroke
Brief Title: Implant for Walking After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Case Western Reserve University (Other); Louis Stokes VA Medical Center (U.S. Federal Agency); Cleveland State University (Other)
Responsible Party: Principal Investigator, Nathaniel Makowski, Assistant Professor, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: StudyID00000125
Record Dates: First submitted 2023-01-18; First posted 2023-02-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hemiplegia; Gait, Hemiplegic
MeSH Terms: conditions — Stroke; Hemiplegia; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Implantation, controller development, and evaluation (Experimental): This phase includes installing the device and setting the individual up for home use, creating advanced controllers for walking and evaluating the effect of the device over several months.
  Interventions: Device: IRS-8; Device: IST 12 & IST 16

INTERVENTIONS:
Device: IRS-8 — Implanted Receiver Stimulator (IRS) delivering 8 channels of stimulation. Appropriate for muscle-based (intramuscular or epimysial) electrodes only
Device: IST 12 & IST 16 — Implantable Stimulator Telemeter (IST) that provides 12 independent channels of stimulation with the option of 2 channels of bipolar myoelectric signal recording, or 16 independent stimulus channels. Suitable for muscle-based or nerve cuff electrodes such as the CWRU Spiral, Flat Interface Nerve Electrode (FINE) or Composite-Flat Interface Nerve Electrode (C-FINE).

SUMMARY:
This is a device study that will evaluate the effect of an implanted stimulator on improving walking in stroke survivors. There are two phases in the study: 1) Screening - this phase determines if the individual is a good candidate to receive an implanted system, 2) Implantation, controller development, and evaluation - this phase includes installing the device and setting the individual up for home use, creating advanced controllers for walking and evaluating the effect of the device over several months.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of neural stimulation for improving walking after stroke. Participants will undergo surgery to implant a stimulator and electrodes to activate muscles used during walking. The device delivers electrical pulses to the nerves causing the muscles to contract to perform functional movements. The system coordinates assistance based on external sensors. After receiving the implanted device, participants undergo training to use the device to assist walking. Evaluations are completed prior to surgery as well after training and at later follow up sessions.

ELIGIBILITY:
Inclusion Criteria:

* At least 6-months post stroke
* Age 21 to 75 years old
* Able to ambulate, but does not require the assistance of more than one person
* Walk slower than 0.8m/s during a 10m walk test
* Lower extremity Fugl-Meyer Motor Assessment (FMA) <= 20
* Reduced peak hip, knee and/or ankle range of motion during stance or swing phases
* Modified Ashworth Scale (MAS) <= 2 at the above joints during passive flexion and extension
* Innervated and excitable lower extremity and trunk musculature
* Appropriate body habitus (height and weight within acceptable limits as determined by study physician)
* Adequate social support and stability
* Willingness to comply with follow-up procedures
* Neurologically stable as determined by a physician

Exclusion Criteria:

* Non-English speaking
* Significant range of motion limitations (lacking hip extension, etc.)
* History of spontaneous fractures or other evidence of excessively low bone density
* Acute orthopedic problems (severe scoliosis, joint dislocations, etc.)
* Medical complications (cardiac abnormalities, skin breakdowns, uncontrolled seizures, immunological/pulmonary/renal/circulatory compromise, additional neurologic conditions etc.)
* Cardiovascular or pulmonary disease
* Uncontrolled diabetes or hypertension
* Presence of a demand pacemaker or cardiac defibrillator
* Pregnancy
* Complications of stroke that result in an increased risk of falls (apraxia, uncompensated hemineglect, hemianopsia etc.)
* Significant history of repeated falls
* Severely impaired cognition and communication
* Any other medical or psychological condition that would be a contraindication

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Gait speed | baseline, ~18 weeks post implant, ~44 week post implant
  The 10mWT is used to assess walking speed in meters/second (m/s) over a short distance.
  Gait speed is how we're evaluating whether the advanced controller works better than a simple generic triggering approach.

SECONDARY OUTCOMES:
Difference in Usability Rating Scale (URS) | baseline, ~18 weeks post implant, ~44-week post implant
  participants will rate the task on a seven-point scale from "very easy" (3) to "very difficult" (-3). Difficulty will be assessed after the 10 m walk test

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Makowski, PhD, Principal Investigator — MetroHealth System, Ohio
Locations (2):
- United States (2):
  - Louis Stokes Cleveland Veterans Affairs Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
De-identified assessment data will be shared via NICHD DASH
Time Frame: Data will become available after study completion
Access Criteria: De-identified data will be available anyone with access to the NICHD DASH repository